CLINICAL TRIAL: NCT02554643
Title: Soccer and Health: Impact of Nutritional Intervention and Recreational Soccer Training in Patients With Type 2 Diabetes Mellitus
Brief Title: Soccer and Health: Diet and Exercise on Type 2 Diabetes Mellitus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Exercise on Type 2 Diabetes
Record Dates: First submitted 2015-09-17; First posted 2015-09-18 (Estimated); Last update posted 2015-09-24 (Estimated); Status verified 2015-09

CONDITIONS: Type 2 Diabetes
Keywords: intermittent exercise; continuous exercise; blood glucose; intramyocellular lipids; diabetes; gene expression
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — Diet; Running

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Diet & Soccer (Experimental): Nutritional Intervention (Diet) once a week, during 12 weeks
  + Soccer training, 3 times a week, during 12 weeks
  Interventions: Other: Diet; Other: Soccer
- Diet & Running (Experimental): Nutritional Intervention (Diet) once a week, during 12 weeks
  + Running training, 3 times a week, during 12 weeks
  Interventions: Other: Diet; Other: Running
- Diet (Active Comparator): Nutritional Intervention (Diet) once a week, during 12 weeks
  Interventions: Other: Soccer; Other: Running

INTERVENTIONS:
Other: Diet — Nutrition intervention, once a week during 12 weeks
  Arms: Diet & Running; Diet & Soccer
Other: Soccer — Nutrition intervention, once a week during 12 weeks + Soccer training, 3 x week, during 12 weeks
  Arms: Diet; Diet & Soccer
Other: Running — Nutrition intervention, once a week during 12 weeks + Running training, 3 x week, during 12 weeks
  Arms: Diet; Diet & Running

SUMMARY:
The present study aims to evaluate the impact of a soccer training program lasting 12 weeks in patients with type 2 diabetes mellitus. 60 sedentary adults and elderly patients with type 2 diabetes mellitus (age: 50-75 y), with a BMI > 25kg/m2 and > 29kg/m2, respectively, from the Hospital of the Medical Faculty of São Paulo University will participate in this study. They will be randomly divided in 3 groups (soccer, running and control). All patients will undergo the following assessments: anthropometric, dietary, physical performance, inflammatory, metabolic and hormonal parameters such as gene expression, bone markers and predictors of cardiovascular disease. In addition the investigators aim to evaluate the body composition of these patients by DXA, and muscle and visceral lipids content by proton spectroscopic MRI.

DETAILED DESCRIPTION:
The present study aims to evaluate the regular soccer practice on cardiorespiratory fitness, body composition, bone health and metabolic and hormonal variables, and compare it with other types of classic aerobic training, such as running, for example .

Soccer is a high popularity team sport, with more than 400 million active practitioners in the world, and due to various motivational and social factors of this activity we can consider it as a great tool potential in promoting the health of sedentary individuals, but football fans. Thus, we believe that the combined use of exercises that make up the soccer training, such as running, walking, sprints, acceleration, deceleration, jumps, side court, dribbling, etc., can result in significant adaptive changes in the physiological system, contributing improvements in cardiovascular function, bone mineralization in muscle strength, physical performance and metabolism of lipids and glucose.

Therefore we aimed to investigate in patients with diabetes mellitus type 2 the impact of a soccer training program with 12 weeks:

* body composition, by examining DXA, assessing the content of lean mass and fat mass;
* the concentration of muscle and visceral fat by means of nuclear magnetic resonance spectroscopy;
* the bone markers for the quantification of osteocalcin hormone, carboxy terminal telopeptides (CTX), propeptide amino-terminal of procollagen type I (P1NP), parathyroid hormone (PTH) and 25-hydroxy vitamin D, growth factor insulin-like-1 free ( IGF1-free);

As a secondary objective, we intend to evaluate the impact of soccer training and classic aerobic exercise on metabolic and hormonal variables of type 2 diabetic patients:

* the parameters of cardiovascular disease, for investigating blood pressure and quantification of lipid fractions (total cholesterol and fractions, triglycerides) and C-reactive protein;
* physical performance, evaluating the physical capacity by examining ergospirometry;
* and the metabolic variables, enzymatic and hormonal following: blood glucose, glycated hemoglobin (HbA1c), tolerance test oral glucose (OGTT), blood lactate, free fatty acids, blood count, insulin, proinsulin, leptin, adiponectin, and enzymes AST, ALT, CK and DHL.

ELIGIBILITY:
Inclusion Criteria: patients with diabetes type 2 diabetes, up to 15 years in duration, HbA1c from 6.5 to 11.0%, with none administration of insulin.

Exclusion Criteria: patients with BMI lower (<) than 25 kg/m2 and higher (>) than 48 kg/m2, blood pressure > 160/100 mm Hg, fasting triglyceride levels of> 500 mg / dL, proteinuria> 100 mg / dL, serum creatinine> 1.5 mg / dL, liver complications, neuropathy or advanced retinopathy, macroangiopathy, diabetic foot, or any other serious health condition that impairs their adherence to the training protocol satisfactorily.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2012-11; Primary Completion 2014-12 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Attenuation of expression of proinflammatory genes verified by qPCR-array technique ranging from at least 5% in pre and post-intervention measurements | 12 weeks

SECONDARY OUTCOMES:
Enhance physical performance verified by oxygen consumption measurement on treadmill | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Maysa Sousa, Principal Investigator — University of Sao Paulo
Locations (1):
- Laboratory of Medical Investigation - LIM 18, University of São Paulo, São Paulo, São Paulo, Brazil